CLINICAL TRIAL: NCT06217588
Title: LCAT Deficiency Disorders: Natural History and Identification of Biomarkers
Brief Title: LCAT (Lecithin Cholesterol Acyl Transferase) Natural History Study
Acronym: LCAT NHS
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 833871
Record Dates: First submitted 2024-01-04; First posted 2024-01-22 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: LCAT Deficiency
Keywords: Renal Disease; LCAT Deficiency; Familial LCAT Deficiency; FLD (Familial LCAT Deficiency); Fish Eye Disease; FED (Fish Eye Disease); Lipoprotein X; LpX (Lipoprotein X); Cardiovascular Disease
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency; Kidney Diseases; Cardiovascular Diseases | interventions — Demography; Genotype

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood (whole blood, PBMC (peripheral blood mononuclear cells), plasma and serum), urine and, when available, histologic samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Demographics, diagnosis type, genotype, lipid profile, renal function profile, treatment allocation, ophthalmology exam, country of residence. — The study will collect extensive historical health data (retrospective), and at baseline will conduct an extensive characterization of the disease progression using the parameters described above.

SUMMARY:
The purpose of the LCAT (Lecithin cholesterol acyl transferase) Natural History Study (LCAT NHS) is to help identify people with a mutation in a gene called LCAT, collect and store information about their medical history and disease course, and to assess for associations and follow changes in clinical features and biomarkers of disease. This information will help health care providers better understand the natural history of disease of LCAT deficiency.

Study staff will collect information from previous clinical visits such as lab tests, physical exam findings, renal and cardiovascular imaging, findings from kidney biopsies and eye exams, and medication and other treatments. As part of this study the investigators are asking participants permission to reach out to their doctors to obtain medical records and stored samples (such as serum or plasma or biopsies) from past visits.

Participants may also be asked to join a web-based patient portal to complete a patient-outcomes survey.

As part of this study, participants will also be asked to do the following things at different times:

* Answer questions about:
* Demographic information (year of birth, age, gender, race/ethnicity, country)
* LCAT deficiency diagnosis such as year of diagnosis, type of diagnosis (clinical, genetic), genotype information/LCAT mutation status
* Medical history and family history and any updates
* A review of medications

If participants are able to come to a study visit in person the following may happen:

Physical examination including vital signs (height, weight, blood pressure, and heart rate) Urine and blood samples for laboratory testing. participants will be required to fast for 10 hours before the blood tests. A small blood sample may also be taken 2-4 hours after a meal.

* The following will be tested: the different types of cholesterol and other fats in the blood (lipids), standard hematology (type and number of blood cells), blood chemistries such as sodium, potassium, and calcium, thyroid function, liver panel (function of the liver), kidney function and the level of protein in urine
* Blood and urine samples may also be stored for future testing
* Genetic material will be collected
* Blood cells may be stored for future research
* Participants will have approximately 4.5 tablespoons of blood drawn annually.
* If not done previously, participants will complete an eye exam.
* Participants may be seen by a doctor specialized in renal disease

ELIGIBILITY:
Inclusion Criteria:

1. Males or Females of any age
2. Subjects with:

   1. a diagnosis of primary LCAT deficiency based on investigator assessment or laboratory results AND/OR
   2. a genetically confirmed mutation in the LCAT gene who are homozygous or compound heterozygous for LCAT loss-of-function mutations
3. Subjects or their legal guardian must be able to comprehend and be willing to provide a signed institutional review board/ethics committee (IRB/EC) approved Informed Consent Form. A waiver of consent will be requested for deceased patients, as determined by local regulatory requirements.

Exclusion Criteria:

1. Secondary causes of LCAT deficiency
2. Any other medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study, or confound the study data

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The registry aims to include data on any patients diagnosed with LCAT deficiency. This includes both patients that have been diagnosed on the basis of genetic analysis and patients that in the opinion of their physician meet the clinical criteria for a diagnosis of LCAT deficiency.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Reaching 40 Patients | Through study completion, an average of 4 years
  Outreach efforts will be made to reach a total of study 40 participants
Mean Age of Diagnosis | Through study completion, an average of 4 years
  The investigators will determine the mean age of diagnosis of LCAT Deficiency
Average time to develop CKD (Chronic Kidney Disease) | Through study completion, an average of 4 years
  The investigators will assess the average time it takes to develop chronic kidney disease

CONTACTS AND LOCATIONS:
Overall Officials: Marina Cuchel, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vitali C, Bajaj A, Nguyen C, Schnall J, Chen J, Stylianou K, Rader DJ, Cuchel M. A systematic review of the natural history and biomarkers of primary lecithin:cholesterol acyltransferase deficiency. J Lipid Res. 2022 Mar;63(3):100169. doi: 10.1016/j.jlr.2022.100169. Epub 2022 Jan 20. PMID 35065092